CLINICAL TRIAL: NCT00256308
Title: A Phase II Study of Adjuvant Chemoradiation With Weekly Oxaliplatin in Patients With High Risk Resected Squamous Cell Carcinoma of the Head and Neck Region
Brief Title: Adjuvant Chemoradiation With Weekly Oxaliplatin in Resected Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Halted prematurely due to slow accrual
Sponsor: University of California, Irvine (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Sai-Hong Ignatius Ou, HS Associate Clinical Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 04-40; 2004-3999 (Other: University of California, Irvine)
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; oxaliplatin; resected squamous cell carcinoma; Eloxatin™
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Oxaliplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxaliplatin (Experimental): Oxaliplatin-70mg/m2 IV over 120 min once a week during radiation. Radiation-200 centigray (cGy) per day - Megavoltage equipment with energy of Cobalt 60 or higher - Daily from Monday to Friday.
  Interventions: Drug: Oxaliplatin; Procedure: Radiation

INTERVENTIONS:
Drug: Oxaliplatin — 70mg/m2 IV over 120 min once a week during radiation
  Other Names: Eloxatin
Procedure: Radiation — 200 cGy/day - Megavoltage equipment with energy of Cobalt 60 or higher - Daily from Monday to Friday

SUMMARY:
Oxaliplatin-containing regimens have been safely and successfully used in combination with concurrent radiation in treatment of solid tumors such as rectal and esophageal cancers. The Lyon R0-04 phase II trial utilized the combination of Oxaliplatin, infusional 5-fluorouracil (5-FU) and radiation in the treatment of rectal cancer. The trial showed a combined preoperative chemoradiotherapy and Oxaliplatin-containing regimen is well tolerated with no increase surgical toxicity. The good response rate observed warrants its use in further clinical trials.

The combination of oxaliplatin, 5-FU, and radiation also have been used in a Phase I/II trial in esophageal cancer. In this particular trial, eligibility included therapeutically naïve esophageal cancer subjects with clinical disease stages II to IV. Initial doses and schedules for cycle 1 consisted of Oxaliplatin 85 mg/m2 on days 1, 15, and 29; continuous infusion of 5-FU 180 mg/m2 for 24 hours for 35 days; and radiation therapy (RT) 1.8 Gy in 28 fractions starting on day 8. At completion of cycle 1, eligible subjects could undergo an operation or begin cycle 2 without RT. Postoperative subjects were eligible for cycle 2. Stage IV subjects were allowed three cycles in the absence of disease progression. 38 subjects were treated (22 stage IV, 16 stage II-III). 38 eligible subjects received therapy: 22 non-invasively staged as IV and 16 non-invasively staged as IV and 16 non-invasively staged as II and III. 36 subjects completed cycle 1, 29 subjects started cycle 2, and 24 subjects completed cycle 2. The combined-modality therapy was well tolerated, but dose limiting toxicity (DLT) prevented Oxaliplatin and 5-FU escalation. No grade 4 hematologic toxicity was noted. Eleven grade 3 and two grade 4 clinical toxicities were noted in eight subjects. After cycle 1, 29 subjects (81%) had no cancer in the esophageal mucosa. 13 subjects underwent an operation with intent to resect the esophagus and 5 subjects (38%) exhibited pathologic complete responses. There was no surgical mortality. Only 1 subject developed post-operative tracheoesphageal fistula. The results of these trials described above indicated that combination of oxaliplatin and radiation is safe and efficacious and dose not compromise surgical wound healing, repair and clinical outcome.

DETAILED DESCRIPTION:
Adjuvant treatment of resected head and neck cancers The incidence of locoregional failures and distant metastasis is high after primary resection of squamous cell carcinoma of the head and neck (HNSCC), especially in patients with unfavorable prognostic factors such as residual disease, histological evidence of extracapsular spread, and/or multiple neck nodes. RT is indicated as an adjuvant therapy to surgery. In the past 2 decades, RT was mainly delivered post-operatively, and the therapeutic gain with this combination is now well documented. Despite an overall 2-year freedom of recurrance of approximately of 70-75%, survival rates are usually poor in the whole HNSCC patient population, and they usually do not exceed 30 to 35% at 5 years. The incidence of metastases in locally advanced but resectable head and neck cancer can reach 15 to 20%. The role of systemic chemotherapy has been tested in clinical trials to determine if the addition of chemotherapy can decrease locoregional and distant failure and improve survival.

Oxaliplatin and radiation in solid tumors Oxalipaltin-containing regimens have been safely and successfully used in combination with concurrent radiation in treatment of solid tumors such as rectal and esophageal cancers. Results of previous trials indicated that combination of oxaliplatin and radiation is safe and efficacious and dose not compromise surgical wound healing, repair and clinical outcome.

Oxaliplatin and radiation in head and neck cancer Oxaliplatin and radiation has been used in a randomized phase II study comparing standard radiation with or without weekly oxaliplatin in the treatment of locally advanced nasopharyngeal carcinoma. Radiation was administered at 70-74 Gy to the primary tumor site, 60-64 Gy to the involved areas of the neck and 50 Gy to the uninvolved area of the neck. Chemotherapy with oxaliplatin at 70 mg/m2 was given weekly for 6 courses with standard radiation in the investigational arm. Interim results concurrent radiation with weekly oxaliplatin resulted in a higher complete response in the primary tumor site and in the cervical lymph nodes. There was no difference in the incidences of dry mouth, stomatitis, skin reaction, peripheral neuropathy or hematological toxicities between the 2 treatment arms. Patients receiving the concurrent radiation and oxaliplatin treatment did experience more gastrointestinal toxicities mostly nausea and vomiting. The only grade 3 toxicities are thrombocytopenia (5.1%), nausea/vomiting (12.8%) and skin reaction (25.6%).

Microscopically involved margins, involvement of two or more nodes, extracapusular spread, presence of perineural involvement, and vascular embolisms are associated with an approximately 25% to 30% probability of developing locoregional failure. The addition of cisplatin to radiation reduces the locoregional failure and distant metastasis. We propose to investigate the toxicities of using weekly oxaliplatin with radiation in the treatment of high risk resected head and neck patients since oxaliplatin has a better side effects profile. The high risk factors will be the same criteria utilized in both RTOG 9501 and EORTC 22931. They include microscopically involved margins, involvement of two or more nodes, extracapusular spread, presence of perineural involvement, vascular embolisms, and oral cavity or oropharyngeal carcinoma with lymph nodes metastasis at level IV or V.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have histologically or cytologically confirmed diagnosis of squamous cell carcinoma of the head and neck region. Primary tumor sites include: oral cavity, pharynx (oropharynx, hypopharynx), or larynx (supraglottis, glottis subglottis). Nasopharynx primary will be excluded.
* The resected tumor must have one or more of the following high risk features: histologic extracapsular nodal extension involvement of ≥ 2 regional lymph nodes, mucosal margin of resection with invasive cancer (limited to microscopic detection only), tumor with perineural invasion, tumor with lymphovascular invasion, oral cavity and oropharynx carcinomas with positive lymph nodes metastasis at level IV or V.
* Radiation must begin within 28 to 56 days after surgical resection.
* All subjects must be 18 years of age or older.
* Subjects must have a Zubrod performance of 0-2.

Exclusion Criteria:

* Subjects must not have distant metastatic disease (M1).
* Subjects must NOT have prior therapy with oxaliplatin.
* Subjects with any evidence of active or uncontrolled infection, recent myocardial infection, unstable angina, or life-threatening arrhythmia are not eligible.
* Patients with severe psychiatric disorder are not eligible.
* No other prior malignancy is allowed except for adequately treated basal cell or squamous cell carcinoma, in situ cervical cancer, or adequately treated Stage I and II cancer from which the patient is in complete remission, or any other malignancy from which the patient has been disease-free for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-02; Primary Completion 2010-05 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sai-Hong Ignatius Ou, MD, PhD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study start date: February 2005 Primary completion date: May 2010 Study completion date: October 2011
Period: Overall Study
Arm/Group | Oxaliplatin
Started | 6
Completed | 4
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Oxaliplatin
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  Caucasian | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Frequency and Severity of Toxicities
Description: Study was terminated by funding source for slow accrual. Upon termination notification, the IRB closure was submitted and all research procedures stopped, inclusive of completing any analysis of data collected.
Time Frame: 2 years
Population: Although data were collected, events were not analyzed at the time of collection for relatedness to treatment and this analysis cannot be performed retrospectively due to lack of access to complete patient records.
Arm/Group | Oxaliplatin
Number analyzed (Participants) | 0

2. Secondary Outcome: Locoregional Control Rate
Description: as for outcome 1
Time Frame: 2 years
Population: Study was terminated by funding source for slow accrual. Upon termination notification, all research procedures stopped, inclusive of completing any analysis of data collected. Specific information about collection of data could not be located.
Arm/Group | Oxaliplatin
Number analyzed (Participants) | 0

3. Secondary Outcome: Disease-free Survival Rate
Description: Study was terminated by funding source for slow accrual. Upon termination notification, the IRB closure was submitted and all research procedures stopped, inclusive of completing any analysis of data collected.
  Progression-free survival: from date of registration to date of first observation of progressive disease, death due to any cause or symptomatic deterioration
  Progression: Appearance of any new lesion/site. The site of the new lesion will be recorded. Death due to disease without prior documentation of progression and without symptomatic deterioration Symptomatic deterioration: Global deterioration of health status requiring discontinuation of treatment without objective evidence of progression. Efforts should be made to obtain objective evidence of progression after discontinuation
Time Frame: 2 years
Population: 4 participants completed survival follow-up. 1 patient had progressive disease and stopped study drug, discovered during follow-up that patient had expired in hospice care. 1 patient completed study treatment but expired in follow up due to staph infection and complications from disease in hospice care.
Measure: Count of Participants; unit: Participants
Arm/Group | Oxaliplatin
Number analyzed (Participants) | 6
Participants
  Disease Free | 4
  Progressive Disease | 1
  Unknown | 1

4. Secondary Outcome: Overall Survival Rate
Description: Study was terminated by funding source for slow accrual. Upon termination notification, the IRB closure was submitted and all research procedures stopped, inclusive of completing any analysis of data collected.
  From date of registration to date of death due to any cause
Time Frame: 2 years
Population: 4 participants completed follow up period. 2 participants expired in the follow up period. 1 due to progressive disease and 1 due to staph infection and secondary cause of death due to disease complications.
Measure: Count of Participants; unit: Participants
Arm/Group | Oxaliplatin
Number analyzed (Participants) | 6
Participants
  Alive | 4
  Deceased | 2

5. Secondary Outcome: Sites of Relapse
Description: as for outcome 1
Time Frame: 2 years
Population: 4 participants completed the study without any signs of disease. Only 1 participant had progressive disease but does not appear to be a relapse. No information provided to indicate whether other expired participant experienced a relapse.
Measure: Count of Participants; unit: Participants
Arm/Group | Oxaliplatin
Number analyzed (Participants) | 6
Participants
  No evidence of Relapse | 5
  Unknown | 1

ADVERSE EVENTS:
Time Frame: 2 years
Description: Known adverse events were reported; however, this may not be a complete representation of the adverse events collected in the study due to limited access to the data.
Arm/Group | Oxaliplatin
All-Cause Mortality (participants affected / at risk) | 2/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin (N=6)
Mucositis (Gastrointestinal disorders) | 1
Dermitis (Skin and subcutaneous tissue disorders) | 1
Dry Mouth (General disorders) | 2 — This adverse event is being reported in this section as a grade determination could not be identified in the patient chart.
Pain (General disorders) | 1 — Due to exposed bone inside of the mouth. This event is being reported in this section as a grade determination could not be identified in the patient chart.
Nausea (General disorders) | 1 — This adverse event is being reported in this section as a grade determination could not be identified in the patient chart.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin (N=6)
Red Skin (Skin and subcutaneous tissue disorders) | 1
Elevated Creatinine (Renal and urinary disorders) | 1
Fever (General disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Hypomagnesemia (Blood and lymphatic system disorders) | 1
Hypertension (Cardiac disorders) | 1
Constipation (Renal and urinary disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Alopecia (Immune system disorders) | 1
Emesis (General disorders) | 1
Sensory Neuropathy (Nervous system disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Pain (General disorders) | 1 — located in mouth
Sensitivity to Cold (General disorders) | 1
Peripheral Neuropathy (Nervous system disorders) | 1
Erythma (Skin and subcutaneous tissue disorders) | 1
Mucositis (General disorders) | 1
Dry Mouth (General disorders) | 1
Weight Loss (General disorders) | 1
Headaches (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes